CLINICAL TRIAL: NCT02587260
Title: Hunting for the Off-Target Properties of Ticagrelor on Endothelial Function and Other Circulating Biomarkers in Humans
Brief Title: Hunting for the Off-Target Properties of Ticagrelor on Endothelial Function in Humans (HI-TECH)
Acronym: HI-TECH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Covance (Industry)
Responsible Party: Principal Investigator, Marco Valgimigli, Coordinating Investigator/Project Leader, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL51124.078.14; 2014-004189-64 (EudraCT Number)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Cardiovascular Diseases
Keywords: P2Y12 inhibitors; Acute Coronary Syndrome (ACS); Endothelial function; Adenosine measurement in human subject; Endopath
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Ticagrelor; Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Latin square design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence I (Active Comparator): Ticagrelor in the period I Prasugrel in the period II Clopidogrel in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel
- Sequence II (Active Comparator): Ticagrelor in the period I Clopidogrel in the period II Prasugrel in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel
- Sequence III (Active Comparator): Prasugrel in the period I Ticagrelor in the period II Clopidogrel in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel
- Sequence IV (Active Comparator): Prasugrel in the period I Clopidogrel in the period II Ticagrelor in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel
- Sequence V (Active Comparator): Clopidogrel in the period I Ticagrelor in the period II Prasugrel in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel
- Sequence VI (Active Comparator): Clopidogrel in the period I Prasugrel in the period II Ticagrelor in the period III
  Interventions: Drug: Ticagrelor; Drug: Prasugrel; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Comparison of ticagrelor with respect to prasugrel and clopidogrel in a different sequence
  Other Names: Brilique
Drug: Prasugrel — Comparison of ticagrelor with respect to prasugrel and clopidogrel in a different sequence
  Other Names: Efient
Drug: Clopidogrel — Comparison of ticagrelor with respect to prasugrel and clopidogrel in a different sequence
  Other Names: Plavix

SUMMARY:
The purpose of this randomized, cross-over study, is to ascertain if ticagrelor, but not prasugrel or clopidogrel, is associated to an improved endothelial function as assessed with peripheral arterial tonometry and markers of endothelial function measurement in post-ACS patients.

DETAILED DESCRIPTION:
Extensive literature documents that endothelial dysfunction is associated with almost every condition predisposing to atherosclerosis and cardiovascular disease. Hence, endothelial dysfunction is significantly associated with the burden of cardiovascular risk and can be considered a barometer of the total risk burden. Importantly, microvascular dysfunction has been shown to increase risk of future cardiovascular events.

This study aims to clarify if ticagrelor, but not prasugrel or clopidogrel is associated to an improved reactive hyperemia index (RHI) and circulating levels of specific biomarkers of endothelial function, at treatment steady state. Ticagrelor has previously been demonstrated to increase adenosine levels by inhibiting adenosine reuptake in red blood cells, by inhibiting the equilibrative nucleoside transporter (ENT)-1. Furthermore, ticagrelor can induce adenosine triphosphate (ATP) release from human red blood cells. Interestingly, ticagrelor, but not clopidogrel or prasugrel have been recently shown to be associated to an improved endothelial function as evaluated with peripheral arterial tonometry after forearm ischemia.

Post-ACS patients (who experienced an acute coronary syndrome and thereby started therapy with an oral P2Y12 inhibitor at least 30 days before) will be consecutively screened for possible inclusion. Patients will then be randomised to receive in a sequential manner the three oral P2Y12 blockers (i.e.) ticagrelor, prasugrel or clopidogrel for at least 30 days each, according to a balanced cross-over study design including the sequences below:

Seq\ Per P.I P.II P.III S.I T P C S.II T C P S.III P T C S.IV P C T S.V C T P S.VI C P T During the three months study period the therapy with the P2Y12 inhibitor will be switched as for randomization sequence scheme.

When started, each drug will be given with the corresponding loading dose of 600 mg for clopidogrel and then continued at 75 mg/day, 180 mg for ticagrelor and then continued at 90 mg b.i.d. and 60 mg for prasugrel and then continued at 10 mg/day (5 mg/day for patients ≥75 years or weighing ≤ 60 kg).

The main measurements, including reactive hypermedia index, PRU, aspirin reaction units, and circulating markers of endothelial function will be performed at baseline, after P2Y12-inhibitor loading dose, before and after P2Y12-inhibitor maintenance dose.

During the visit, blood pressure will be measured in the contralateral arm before examination. The EndoPAT probes will be placed on the index fingers. If the index finger will be missing or deformed, another finger will be used, using the same finger on both hands. Baseline registration will be conducted for 5 min. The test arm will be then occluded for 5 min, using a standard blood pressure cuff placed on the upper arm. Subsequently, the cuff was deflated and the registration continued for 5 more minutes. After EndoPAT, blood will be drawn to collect serum and plasma for biomarkers assessment [Asymmetrical dimethylarginine (ADMA), adenosine plasma concentration, von willebrand factor antigen, endothelin-1, C-reactive protein, soluble fms-like tyrosine kinase-1 (sFLT-1), intercellular cell adhesion molecule-1 (ICAM-1), vascular cell adhesion molecule-1 (VCAM-1), prothrombin fragment 1+2, fibrinopeptide A, and thrombin-antithrombin complex (TAT)]. To assess the relationship between residual platelet reactivity or percent inhibition and effect of P2Y12 oral blocker on endothelial function, platelet function testing will be also carried out acutely and at treatment steady state by means of the Verifynow system using both P2Y12 and aspirin assays.

Based on previous findings, we set mean RHI at 1.8 with a within subjects SD of 0.31. Hence, 36 patients completing all sequences (i.e. 6 pt/sequence) will provide 90% power to detect a 10% RHI relative change in the ticagrelor group with a two-sided alpha level at 5%. To account for drop outs as well as incomplete data assessment at all time points, a final sample size of 50 patients will be recruited.

Patients will be provided with a regular drug prescription (standard of care medication). At each follow-up the investigator will collect information about adherence to the study drug and register the charge number of the prescribed P2Y12.

Allocation of study treatment will be performed via a web-based interactive randomization system, based on a computer-generated random sequence with a random block size stratified according to the type of P2Y12 inhibitor (ticagrelor vs prasugrel vs clopidogrel) as well as for the presence of diabetes mellitus.

Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to study. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded. Serious adverse events in this study are considered to be extremely rare.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients who experienced an Acute Coronary Syndrome (including STEMI or NSTEMI) at least 30 days before.
* Patients on ongoing treatment for at least 30 days with dual anti-platelet therapy consisting of aspirin, at doses of 75-160 mg daily and one commercially available P2Y12 oral inhibitor , including ticagrelor, clopidogrel or prasugrel.
* Patients who remained free from bleeding (defined as BARC type 2 or greater) or ischemic recurrences.
* Signed informed consent All inclusion criteria are required.

Exclusion Criteria:

* Administration of fibrinolytics or glycoprotein IIb/IIIa inhibitors in the previous 30 days.
* Major surgery within 30 days or any planned surgical or percutaneous intervention.
* Active bleeding or previous clinical relevant bleeding or stroke in the last 6 months.
* Previous transient ischemic attack or intracranial bleeding.
* Thrombocytopenia.
* Oral anticoagulant therapy.
* Vasculitis or any know immunological disorder.
* Severe hepatic failure.
* Uncontrolled hypertension (systolic or diastolic arterial pressure >180 mmHg or 120, respectively, despite medical therapy).
* Known intolerance to aspirin or to clopidogrel or prasugrel or ticagrelor.
* Limited life expectancy, e.g. neoplasms, others.
* Inability to obtain informed consent.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Improvement of endothelial function at steady state | After 30 days of therapy with assigned P2Y12-inhibitor
  Evaluation if ticagrelor, at steady state (i.e. after 30 day therapy), will be associated to an improved endothelial function as compared to clopidogrel or prasugrel when assessed with endopath system 1-2 hour(s) after maintenance drug intake.

SECONDARY OUTCOMES:
Improvement of endothelial function, both acutely and at steady state | One or 2 hour(s) after P2Y12-inhibitor loading dose administration and before and 1 or 2 hour(s) after maintenance dose administration
  To assess if treatment with ticagrelor, both acutely and at steady state is associated to an improved endothelial function phenotype as compared to clopidogrel or prasugrel. The assessment is made with measurement of blood markers of endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Policlinico San Matteo, Pavia, Italy
- Netherlands (2):
  - VU Medical Center, Amsterdam
  - Erasmus MC, Rotterdam
- Hospital Clinic, Barcelona, Spain
- Inselspitäl University Medical Center, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hochberg Y, Benjamini Y. More powerful procedures for multiple significance testing. Stat Med. 1990 Jul;9(7):811-8. doi: 10.1002/sim.4780090710. PMID 2218183
- [Result] Flammer AJ, Anderson T, Celermajer DS, Creager MA, Deanfield J, Ganz P, Hamburg NM, Luscher TF, Shechter M, Taddei S, Vita JA, Lerman A. The assessment of endothelial function: from research into clinical practice. Circulation. 2012 Aug 7;126(6):753-67. doi: 10.1161/CIRCULATIONAHA.112.093245. PMID 22869857
- [Result] Cattaneo M, Schulz R, Nylander S. Adenosine-mediated effects of ticagrelor: evidence and potential clinical relevance. J Am Coll Cardiol. 2014 Jun 17;63(23):2503-2509. doi: 10.1016/j.jacc.2014.03.031. Epub 2014 Apr 23. PMID 24768873
- [Result] Bonello L, Laine M, Kipson N, Mancini J, Helal O, Fromonot J, Gariboldi V, Condo J, Thuny F, Frere C, Camoin-Jau L, Paganelli F, Dignat-George F, Guieu R. Ticagrelor increases adenosine plasma concentration in patients with an acute coronary syndrome. J Am Coll Cardiol. 2014 Mar 11;63(9):872-7. doi: 10.1016/j.jacc.2013.09.067. Epub 2013 Nov 27. PMID 24291273
- [Result] Torngren K, Ohman J, Salmi H, Larsson J, Erlinge D. Ticagrelor improves peripheral arterial function in patients with a previous acute coronary syndrome. Cardiology. 2013;124(4):252-8. doi: 10.1159/000347122. Epub 2013 Apr 9. PMID 23594617
- [Result] McCrea CE, Skulas-Ray AC, Chow M, West SG. Test-retest reliability of pulse amplitude tonometry measures of vascular endothelial function: implications for clinical trial design. Vasc Med. 2012 Feb;17(1):29-36. doi: 10.1177/1358863X11433188. PMID 22363016
- [Derived] Ariotti S, Ortega-Paz L, van Leeuwen M, Brugaletta S, Leonardi S, Akkerhuis KM, Rimoldi SF, Janssens G, Gianni U, van den Berge JC, Karagiannis A, Windecker S, Valgimigli M; HI-TECH Investigators. Effects of Ticagrelor, Prasugrel, or Clopidogrel on Endothelial Function and Other Vascular Biomarkers: A Randomized Crossover Study. JACC Cardiovasc Interv. 2018 Aug 27;11(16):1576-1586. doi: 10.1016/j.jcin.2018.04.022. Epub 2018 May 24. PMID 29805112
- [Derived] Ariotti S, van Leeuwen M, Brugaletta S, Leonardi S, Akkerhuis KM, Rimoldi SF, Janssens GN, Ortega-Paz L, Gianni U, van den Berge JC, Karagiannis A, Windecker S, Valgimigli M; HI-TECH Investigators. Effects of Ticagrelor, Prasugrel, or Clopidogrel at Steady State on Endothelial Function. J Am Coll Cardiol. 2018 Mar 20;71(11):1289-1291. doi: 10.1016/j.jacc.2018.01.027. No abstract available. PMID 29544613